CLINICAL TRIAL: NCT06088407
Title: Tranexamic Acid Prophylaxis for Heterotopic Ossification in Elbow Fracture-Dislocation Surgery: A Prospective Randomized Trial
Brief Title: Tranexamic Acid Prophylaxis for Heterotopic Ossification in Elbow Fracture-Dislocation Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0052-16-ASF
Record Dates: First submitted 2023-09-26; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Elbow Dislocation; Heterotopic Ossification
MeSH Terms: conditions — Ossification, Heterotopic | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- With tranexamic acid (Experimental): Patient undergoing surgery for elbow fracture-dislocation randomized to be treated with tranexamic acid intraoperatively.
  The patients received intravenous 1 gram tranexamic acid in 100ml normal saline 30 minutes before skin incision and a second dose of intravenous 1 gram tranexamic acid in 100 ml of normal saline during wound closure.
  Interventions: Drug: with Tranexamic acid
- Without tranexamic acid (No Intervention): Patient undergoing surgery for elbow fracture-dislocation randomized to be treated without tranexamic acid intraoperatively

INTERVENTIONS:
Drug: with Tranexamic acid — Patients undergoing surgery for elbow fracture-dislocation randomized to be treated with tranexamic acid intravenous intraoperatively
  Arms: With tranexamic acid

SUMMARY:
Heterotopic ossification (HO) following elbow fracture-dislocation is a well-recognized condition that can lead to reduced range of motion, increased pain, and the necessity for repeat surgeries.

Inflammation serves as a pivotal initiating factor in the formation of (HO) following a traumatic event. The inflammatory cascade triggered can lead to the dysregulation of tissue homeostasis, thereby promoting the aberrant formation of ectopic bone. Tranexamic acid (TXA), a Food and Drug Administration (FDA) approved synthetic antifibrinolytic agent, has garnered significant attention for its potential to mitigate the inflammatory response in the context of orthopaedic surgical procedures.

This study aims to investigate the hypothesis that reducing soft tissue hematoma during elbow fracture-dislocation surgery through the intraoperative administration of TXA, can alleviate the occurrence or severity of ectopic bone formation.

Methods: A prospective randomized study was conducted on patients with elbow fracture-dislocation who underwent surgery between 2016 and 2022. A total of 50 patients were enrolled and randomly assigned to two groups. The first group received 1 gram of intravenous tranexamic acid before the operation, followed by an additional 1 gram intravenously during wound closure. The second group did not receive any anti-bleeding medication. Patients were followed up at intervals of 2 weeks, 6 weeks, 3 months, and as needed after the surgery. At the end of the follow-up period, there were 23 patients in the first group and 24 in the second group, with a median follow-up duration of 12.7 months. All patients did not receive any other form of HO prophylaxis. Postoperative radiographs and clinical outcomes were assessed and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. traumatic non-pathological elbow fracture-dislocation.
2. age 18 years or older.
3. presentation within 2 weeks of injury.
4. Willingness to participate in the study

Exclusion Criteria:

1. Inability to provide consent for research participation.
2. Active infection in the operated limb.
3. Previous hip fracture.
4. Head injury.
5. History of deep vein thrombosis (DVT).
6. History of venous thromboembolism (VTE).
7. Ischemic heart event within the last six months.
8. Stroke (CVA) within the last six months.
9. Coagulopathies.
10. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02-21 (Actual); Primary Completion 2023-09-03 (Actual); Study Completion 2023-09-03 (Actual)

PRIMARY OUTCOMES:
Presence of Heterotopic Ossification in plain radiographs | 2 weeks- 1 year
  Heterotopic Ossification presence, defined as new bone formation that had not been present in the imaging studies made at the time of the injury

SECONDARY OUTCOMES:
Functional elbow Range of motion assessment | 2 weeks - 1 year
  Elbow range of motion throughout the follow-up. The range of motion of the elbow was evaluated in degrees using a full circle goniometer (Jamar, Duluth, Minnesota, United States). Functional range of motion was classified as 30-130 degrees of extension-flexion according to the description by Morrey et al (A biomechanical study of normal functional elbow motion. B F Morrey, L J Askew, E Y Chao. J Bone Joint Surg Am. 1981 Jul;63(6):872-7.). Patients with worse range of motion then 30-130 degrees (larger then 30 degrees extension and lower then 130 degrees of flexion) were classified as patients with non-functional elbow range of motion.
Heterotopic Ossification Classification System Score | 2 weeks - 1 year
  Heterotopic Ossification Classification System by Hastings and Graham (The classification and treatment of heterotopic ossification about the elbow and forearm. H Hastings 2nd, T J Graham. Hand Clin. 1994 Aug;10(3):417-37.).
  The score is between I-III, where I means radiographic heterotopic ossification without elbow motion limitations (better outcome) and III means radiographic heterotopic ossification with no elbow motion (worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofeh Medical Center (Yitzhak Shamir Medical Center), Be’er Ya‘aqov, Israel